CLINICAL TRIAL: NCT00055692
Title: Bevacizumab (RhuMAB-VEGF) In Hepatocellular Cancer For Patients With Unresectable Tumor (Without Invasion Of The Main Portal Vein Or Metastatic Disease) A Phase II Study
Brief Title: Bevacizumab in Treating Patients With Unresectable Nonmetastatic Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02518; NCI-2012-02518 (Other: CTRP (Clinical Trial Reporting Program)); NCI-5611 (Other: NCI/CTEP); 5611 (Other: CTEP); P30CA013330 (NIH); N01CM62204 (NIH); N01CM62203 (NIH)
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2012-12

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (bevacizumab) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1. Treatment continues every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab

INTERVENTIONS:
Biological: bevacizumab — Given orally
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF

SUMMARY:
This phase II trial is to see if bevacizumab works in treating patients who have unresectable nonmetastatic liver cancer that has not spread to the main portal vein. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the efficacy of bevacizumab, in terms of progression-free survival and disease stability and response, in patients with unresectable nonmetastatic hepatocellular cancer (HCC) without main portal vein invasion.

II. Determine the safety of this drug in these patients. III. Assess tumor vascular perfusion kinetics, by dynamic gadolinium-enhanced MRI, in patients before and after treatment with this regimen.

IV. Determine the effect of vascular endothelial growth factor (VEGF)-inhibition by this drug on circulating levels of VEGF and related cytokines that also contribute to HCC pathogenesis (including bFGF, TGF-alpha, and IGF-II) and on potential alterations of these levels on prognostic variables in these patients.

V. Determine the effect of VEGF-inhibition by this drug on hepatic function and hepatitis viral activity in cirrhosis in these patients.

OUTLINE: This is a multicenter, pilot study.

Patients receive bevacizumab IV over 30-90 minutes on day 1. Treatment continues every 2 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 18-46 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed hepatocellular carcinoma

  * Confirmed by needle aspirate, biopsy, or prior surgical resection specimen
* Clinically confirmed hepatocellular carcinoma defined as follows:

  * Cirrhosis or chronic hepatitis B or C virus infection, with 1 or more hypervascular liver masses more than 2 cm
  * Alpha-fetoprotein (AFP) greater than 400 ng/mL OR greater than 3 times normal and doubling in value during the past 3 months
* Deemed unresectable

  * Prior surgical resection allowed
  * Recurrence after hepatic resection or other procedure allowed
  * Tumor that extends into branches of the portal or hepatic veins allowed
  * No tumor invading the main portal vein (portal trunk) or inferior vena cava
  * No tumor occupying more than 50% of the liver volume
* Enlargement/involvement of regional lymph nodes allowed
* At least 1 unidimensionally measurable lesion at least 20 mm

  * No poorly defined lesions
  * No vague hypervascular patches
* Child-Pugh class A or compensated Child-Pugh class B liver dysfunction

  * No Child-Pugh class C or uncompensated class B indicated by active encephalopathy, persistent ascites, or prothrombin time greater than 1.5 times normal
  * Prior ascites allowed if manageable with diuretics alone
  * No repeated paracentesis (more than 1 per month)
* No extrahepatic metastasis
* No documented brain metastases
* No history or clinical evidence of CNS disease (e.g., primary brain tumor, seizures uncontrolled with standard medical therapy, or history of stroke)
* Performance status - ECOG 0-2
* Absolute neutrophil count greater than 1,500/mm^3
* Hemoglobin at least 8 g/dL
* Platelet count at least 75,000/mm^3
* No prior serious bleeding event (unrelated to liver disease)
* No bleeding diathesis
* No coagulopathy
* Bilirubin no greater than 3 mg/dL
* Transaminases less than 5 times upper limit of normal (ULN)
* Albumin at least 2.5 mg/dL
* PTT less than 4 seconds above ULN
* INR less than 1.5 (for patients receiving warfarin)
* Creatinine less than 1.5 g/dL
* Urine protein less than 500 mg/24hrs*

Exclusion criteria:

* No thromboembolic event within the past 12 months
* No clinically significant cardiovascular disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring parenteral antibiotics
* No serious non-healing wound/ulcer or bone fracture
* No variceal bleeding within the past 6 months
* No malignancy within the past 5 years except localized nonmelanoma skin cancer
* No ongoing psychiatric or social situation that would preclude study compliance
* No known hypersensitivity to Chinese hamster ovary cell products
* No known hypersensitivity to other recombinant human antibodies
* No more than 1 prior biologic therapy
* No concurrent interferon
* No concurrent interleukin-2
* No more than 1 prior antineoplastic chemotherapy
* At least 4 weeks since prior invasive surgery, including open biopsy
* At least 2 weeks since prior needle biopsy (core or fine-needle aspirate)
* No concurrent hepatic transplant
* At least 4 weeks since prior anticancer therapy
* No concurrent platelet-stimulating factors (e.g., oprelvekin)
* No concurrent full-dose anticoagulants or thrombolytic agents (except as required to maintain patency of pre-existing, permanent indwelling IV catheters)
* No chronic daily antiplatelet drugs (e.g., aspirin doses of 325 mg/day or higher or non-steroidal anti-inflammatory drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-02; Primary Completion 2008-01 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abby Siegel, Principal Investigator — Montefiore Medical Center - Moses Campus
Locations (1):
- Montefiore Medical Center - Moses Campus, The Bronx, New York, United States

REFERENCES:
- [Result] Siegel AB, Cohen EI, Ocean A, Lehrer D, Goldenberg A, Knox JJ, Chen H, Clark-Garvey S, Weinberg A, Mandeli J, Christos P, Mazumdar M, Popa E, Brown RS Jr, Rafii S, Schwartz JD. Phase II trial evaluating the clinical and biologic effects of bevacizumab in unresectable hepatocellular carcinoma. J Clin Oncol. 2008 Jun 20;26(18):2992-8. doi: 10.1200/JCO.2007.15.9947. PMID 18565886

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 46 patients were enrolled between February 2003 and September 2006
Period: Overall Study
Arm/Group | Treatment (Bevacizumab)
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 58 [21 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 38
Race/Ethnicity, Customized [Number; unit: participants]
  White | 25
  Black | 2
  Hispanic | 5
  Asian | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Time Frame: At 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 46
percentage of participants | 65 [51 to 79]

2. Primary Outcome: Disease Response
Description: MRI scan is required at weeks 8, 16 and then every 12 weeks until disease progression. Per Response Evaluation Criteria in Solid Tumors (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: MRI is required at weeks 8, 16 and then every 12 weeks until disease progression
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 46
participants | 6 [3 to 23]

3. Primary Outcome: Mean Arterial Enhancement, Per Lesion, as Determined by Dynamic Gadolinium-enhanced Magnetic Resonance Imaging (MRI), Before and Following Bevacizumab Therapy.
Time Frame: Baseline and 8 weeks after bevacizumab therapy
Population: Eight consecutive patients enrolled at one site were evaluated before and at 8 weeks after bevacizumab therapy with DCE-MRI.
Measure: Mean (Standard Deviation); unit: relative MR units
Groups:
- Treatment (Bevacizumab): Baseline; Treatment (Bevacizumab): 8 Weeks: Patients receive bevacizumab IV over 30-90 minutes on day 1. Treatment continues every 2 weeks in the absence of disease progression or unacceptable toxicity.
  bevacizumab: Given orally
Arm/Group | Treatment (Bevacizumab): Baseline | Treatment (Bevacizumab): 8 Weeks
Number analyzed (Participants) | 8 | 8
relative MR units | 37.3 (18.4) | 18.4 (12.4)

4. Primary Outcome: Assessment on Circulating Levels of VEGF Which Also Contribute to HCC Pathogenesis and on Potential Alterations of These Levels in the Setting of VEGF-inhibition
Time Frame: During treatment
Population: Six of eight patients were analyzed after 8 weeks of bevacizumab therapy
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 6
pg/mL | 249 (175)

5. Primary Outcome: To Collect Information on Hepatic Function and Hepatitis Viral Activity in Cirrhosis and Upon Potential Alterations in the Setting of VEGF-inhibition
Time Frame: During and after treatment
Population: No data was collected by the principal investigator for this outcome
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Disease Stability
Time Frame: At 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Treatment (Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 22/46
Other Adverse Events (participants affected / at risk) | 41/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bevacizumab) (N=46)
Hypertension (Vascular disorders) | 7 (7)
Proteinuria (Renal and urinary disorders) | 2 (2)
Hemorrhage (Gastrointestinal disorders) | 5 (5)
Arterial thrombosis (Vascular disorders) | 2 (2)
Venous thrombosis (Vascular disorders) | 1 (1)
Increased AST (Investigations) | 1 (1)
Increased ALT (Investigations) | 1 (1)
Increased alkaline phosphatase (Investigations) | 1 (1)
Increased bilirubin (Investigations) | 5 (5)
Ascites (Gastrointestinal disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bevacizumab) (N=46)
Hypertension (Vascular disorders) | 8 (8)
Proteinuria (Renal and urinary disorders) | 17 (17)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hemorrhage (Gastrointestinal disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Thrombocytopenia (Investigations) | 6 (6)
Increased AST (Investigations) | 9 (9)
Increased ALT (Investigations) | 8 (8)
Increased alkaline phosphatase (Investigations) | 4 (4)
Increased bilirubin (Investigations) | 7 (7)
Ascites (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 15 (15)
vomiting (Gastrointestinal disorders) | 5 (5)
Anorexia (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less